CLINICAL TRIAL: NCT01245088
Title: A Pilot Study of Chondroitin Sulfate (CS) for the Treatment of Mild to Moderate Crohn's Disease
Brief Title: Chondroitin Sulfate for Crohn's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support after no patients enrolled
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jeffry A. Katz, Associate Professor of Medicine, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCDZ
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; chondroitin sulfate
MeSH Terms: conditions — Crohn Disease | interventions — Chondroitin Sulfates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chondroitin sulfate (Experimental): 400 mg (one table) TID
  Interventions: Drug: chondroitin sulfate

INTERVENTIONS:
Drug: chondroitin sulfate — 400 mg orally three times daily for 8 weeks

SUMMARY:
Pilot trial of open-label chondroitin sulfate 400 mg TID for adult patients with mild to moderate Crohn's disease. Primary endpoint with be evidence of bilogic effect assessed through serum and tissue cytokine analysis. Secondary endpoints are evidence of clinical effect, endoscopic healing, and histologic improvment. Trial duration is 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Colonic or ileocolonic CD diagnosed for at least 3 months. 2. Active CD, defined as a Crohn's Disease Activity Index (CDAI; Appendix A) [Best 1976] of greater than 200 but less than 320 at the time entry into the study.

  3. Age > 18 years. 4. Patients receiving oral or topical 5-aminosalicylates must be on a stable dose for four weeks prior to enrollment.

  5. Patients on azathioprine, 6-mercaptopurine, or methotrexate must be on stable doses for 14 weeks prior to enrollment.

  6. Patients on corticosteroids must be on stable doses for 2 weeks prior to enrollment.

  7. Patients receiving corticosteroid enemas must be on a stable dose for 3 weeks prior to enrollment.

  8. Patient on biologic therapy with infliximab, adalimumab, or certolizumab must be on stable therapy for 12 weeks prior to enrollment 9. Patient must sign informed consent.

Exclusion Criteria:

* 1. Patients with only small bowel CD, fistulizing CD, or gastroduodenal CD without colonic involvement.

  2. Patients with known ulcerative colitis. 3. Patients expected to require surgery within 30 days for complications of CD. 4. Patients with CD and an intraabdominal abscess. 5. Patients requiring continuous antibiotics; antibiotics may be taken up to the point of enrollment into the study.

  6. Patients with severe cardiac, pulmonary, or renal disease. 7. Patients with a h/o malignancy other than resected basal cell carcinoma of the skin 8. Patients who have participated in another clinical research study in the past 8 weeks.

  9. Patients who are pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Biologic effect on inflammation | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case medical Center, Cleveland, Ohio, United States